CLINICAL TRIAL: NCT02633904
Title: Investigation of the Value of Femoral Shortening Osteotomy During Open Treatment of Developmental Dislocation of the Hip in Waliking Age Group
Brief Title: Investigation of the Femoral Shortening Osteotomy in the Developmental Dislocation of the Hip (FSODDH)
Acronym: FSODDH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: He Jin Peng (Other)
Collaborators: Hunan Children's Hospital (Other Government); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Guangzhou Women and Children's Medical Center (Other); Wuhan Women and Children's Medical Center (Other); Shenzhen Children's Hospital (Other Government); Foshan Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor-Investigator, He Jin Peng, Resident doctor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FSODDH; He Jin Peng (Registry Identifier: Tongji Hospital)
Record Dates: First submitted 2015-12-10; First posted 2015-12-17 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: Hip Dislocation; Femur Head Necrosis
Keywords: Hip Dislocation; Congenital; osteotomy; Femur Head Necrosis
MeSH Terms: conditions — Hip Dislocation; Femur Head Necrosis | interventions — Osteotomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Osteotomy (Active Comparator): Femoral osteotomy are applied in the open treatment of Developmental Dislocation of the Hip （DDH）.
  Interventions: Procedure: Osteotomy
- Non-osteotomy (Experimental): Femoral osteotomy are not applied in the open treatment of Developmental Dislocation of the Hip （DDH）.
  Interventions: Procedure: Non-osteotomy

INTERVENTIONS:
Procedure: Osteotomy — Femoral osteotomy are applied in the open treatment of Developmental Dislocation of the Hip （DDH）.
  Arms: Osteotomy
Procedure: Non-osteotomy — Femoral osteotomy are not applied in the open treatment of Developmental Dislocation of the Hip （DDH）.
  Arms: Non-osteotomy

SUMMARY:
Although older children and high dislocations may be more likely to require a femoral shortening osteotomy, the ultimate decision about whether or not to shorten a given femur should depend on the ease of femoral head reduction in that specific patient. Adding a femoral shortening procedure increases operating time and blood loss, adds a second incision, and necessitates future hardware removal. In addition, an unnecessary femoral shortening osteotomy could overly decrease the soft tissue tension around the joint, putting the hip at risk for redislocation. This study was designed to explore an algorithm based on strict age and radiographic criteria that identify those without the need of femoral osteotomy.

DETAILED DESCRIPTION:
Developmental dislocation of the hip (DDH) is a common disease in children, and its incidence in China is about 9 ‰.There are many different methods in the treatment of DDH. Although older children and high dislocations may be more likely to require a femoral shortening osteotomy, the ultimate decision about whether or not to shorten a given femur should depend on the ease of femoral head reduction in that specific patient. Adding a femoral shortening procedure increases operating time and blood loss, adds a second incision, and necessitates future hardware removal. In addition, an unnecessary femoral shortening osteotomy could overly decrease the soft tissue tension around the joint, putting the hip at risk for redislocation. This study was designed to explore an algorithm based on strict age and radiographic criteria that identify those without the need of femoral osteotomy. From the investigators'clinical experiences and the published papers, younger patients (<24 month of age) and low dislocations (Tonnis level I or II) were more likely to avoid a femoral shortening osteotomy.

ELIGIBILITY:
Inclusion Criteria:

1. Unilateral DDH,age 18-24month.
2. Tonnis degree I or II.
3. Not receive any open treatment.

Exclusion Criteria:

1. Teratologic hip dislocations,
2. Patients with mental, neurological disorders (such as hypoxic-ischemic encephalopathy, epilepsy and dementia) or significant barriers to growth, cerebral palsy, multiple joint contractures disease, dysfunction of liver and kidney , blood disorders, immune deficiency disease and ECG abnormalities.
3. Any children with prior hip surgery were excluded from the series.
4. Parents refused further treatment.

Ages: 18 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2015-12; Primary Completion 2018-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Femur Head Necrosis | 2 years
  Radiological evaluation was performed using standard anterior-posterior radiographs of the pelvis. The presence and grade of femur head necrosis was evaluated according to the method presented by Bucholz and Odgen.
Redislocation | 2 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0.
Acetabular index | 2 years
  Standardized radiographs have been traditionally used in the surveillance of hip dysplasia by measuring the acetabular index, which is the angle subtended between the Hilgenreiner line and a line drawn from the triradiate cartilage to the lateral edge of the acetabulum.

SECONDARY OUTCOMES:
Duration of operation | 1 month
  The time during the operation measured by minute.
Blood loss | 1 month
  The blood lost during the operation measured by milliliter.
Cost | 1 month
  The cost of hospitalization.
Hospital stays | 1 month
  The days stayed in hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Fan J Shao, Doctor, Study Director — Affiliated Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology

IPD SHARING:
Plan to Share IPD: Yes
The single-center data will be published in the form of case-control study.

REFERENCES:
- [Result] Sankar WN, Tang EY, Moseley CF. Predictors of the need for femoral shortening osteotomy during open treatment of developmental dislocation of the hip. J Pediatr Orthop. 2009 Dec;29(8):868-71. doi: 10.1097/BPO.0b013e3181c29cb2. PMID 19934701
- [Result] Pospischill R, Weninger J, Ganger R, Altenhuber J, Grill F. Does open reduction of the developmental dislocated hip increase the risk of osteonecrosis? Clin Orthop Relat Res. 2012 Jan;470(1):250-60. doi: 10.1007/s11999-011-1929-4. Epub 2011 Jun 4. PMID 21643924